CLINICAL TRIAL: NCT04787406
Title: The Effect of Single Session Transcranial Direct Current Stimulation on Sequential Motor Learning in Parkinson's Disease
Brief Title: Motor Learning and tDCS in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20181226002
Record Dates: First submitted 2021-03-01; First posted 2021-03-08 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Transcranial direct current stimulation; Motor sequence learning
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anodal tDCS (Active Comparator): Anodal electrode (35 cm2 sponge electrode) placed over C3. Cathodal electrode (35 cm2 sponge electrode) placed over the right supraorbital area. 20 minutes of stimulation at 2 mA with a 30-second phase-in and phase-out period.
  Interventions: Device: Transcranial direct current stimulation
- Cathodal tDCS (Active Comparator): Cathodal electrode (35 cm2 sponge electrode) placed over C3. Anodal electrode (35 cm2 sponge electrode) placed over the right supraorbital area. 20 minutes of stimulation at 2 mA with a 30-second phase-in and phase-out period.
  Interventions: Device: Transcranial direct current stimulation
- Sham tDCS (Sham Comparator): Anodal electrode (35 cm2 sponge electrode) placed over C3. Cathodal electrode (35 cm2 sponge electrode) placed over the right supraorbital area. Stimulation was phased in for 30 seconds up to 2 mA and then switched off. Stimulation was again phased in for 30 seconds following 20 minutes of no stimulation.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Transcranial electrical stimulation device. A weak direct electrical current, up to 2 mA, is passed between two electrodes placed on the scalp. Electrodes are housed in 35 cm2 sponges saturated with 4 ml of saline solution (0.9 % NaCl) per side, per pad.
  Stimulation is phased in with a 30 second ramp up period prior to the specified stimulation period and phased-out with a ramp down of the current following the specified stimulation period. For sham stimulation, the ramp-up and ramp-down periods are retained, but stimulation is switched off for during the specified stimulation period.
  Other Names: tDCS

SUMMARY:
The present study sought to examine the efficacy of single session transcranial direct current stimulation applied over the primary motor cortex in people with Parkinson's disease on sequential motor learning performance.

DETAILED DESCRIPTION:
Parkinson's disease is characterised by deficits of motor control triggered by impaired basal ganglia function, such as bradykinesia and tremor. Beyond the visibly recognisable motor symptoms of Parkinson's disease, the ability to learn a sequence of movements is also compromised and poses a significant barrier to effective rehabilitation. In healthy individuals, transcranial direct current stimulation applied over the primary motor cortex during motor task practice has been shown to significantly improve motor learning compared to placebo conditions. The present study sought to examine the effect of a single session of transcranial direct current stimulation applied over the primary motor cortex in people with Parkinson's disease on sequential motor learning performance. Participants learnt two finger tapping sequences, with task difficulty indexed by sequence length, and task consolidation further examined using a dual-task paradigm. Task related cortical haemodynamic activity was recorded using functional near-infrared spectroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed (Edinburgh Handedness Inventory; ≥50)
* Cognitively capable (Montreal Cognitive Assessment (MoCA); ≥23)
* Mild to moderate Parkinson's disease severity (Hoehn and Yar disease stage 2-3)

Exclusion Criteria:

* History of stroke
* Comorbidity
* Cephalic implants

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline sequential finger tapping performance | Two assessments: Baseline / pre-intervention, and immediately post-intervention
  A skill index reflecting the accuracy and speed of which participants perform a specified finger tapping sequence.
Change from baseline oxygenated haemoglobin response | Two assessments: Baseline / pre-intervention, and immediately post-intervention
  Task related changes of oxygenated haemoglobin as measured using functional near-infrared spectroscopy.
Change from baseline shape-counting error | Two assessments: Baseline / pre-intervention, and immediately post-intervention
  The percentage of shape counting error during dual task assessments. Sequential finger tapping + visual shape counting task.

CONTACTS AND LOCATIONS:
Overall Officials: Magaret Mak, Dr, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hung Hom, Hong Kong

IPD SHARING:
Plan to Share IPD: No